CLINICAL TRIAL: NCT02120963
Title: The Effect of Person-centered Physical Therapy on Fatigue Related Variables in Persons With Rheumatoid Arthritis- Randomized Controlled Trial
Brief Title: Fatigue in People With Rheumatoid Arthritis- Randomized Controlled Trial
Acronym: RAFatigueRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FatigueRA-RCT
Record Dates: First submitted 2014-01-15; First posted 2014-04-23 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Fatigue; Rheumatoid Arthritis
Keywords: Fatigue; Rheumatoid Arthritis; Physical Therapy; Person-Centred Care
MeSH Terms: conditions — Fatigue; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention program (Experimental): Person-centered physical therapy intervention program
  Interventions: Behavioral: Person-centered physical therapy intervention program
- Control group (No Intervention): Health care as usual

INTERVENTIONS:
Behavioral: Person-centered physical therapy intervention program — Comparison of person-centered physical therapy and control group
  Arms: intervention program

SUMMARY:
Aim: To study if a person-centered physical therapy intervention program contributes to diminished fatigue in people with Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
The effect of person-centered physical therapy on fatigue related variables in peoples with Rheumatoid Arthritis- Randomized controlled trial Aim: To study if a person-centered physical therapy intervention program contributes to diminished fatigue in people with RA.

Hypothesis: That the person-centered treatment program diminishes fatigue and its consequences on daily life.

Design: A controlled randomized interventional trial, assessing effectiveness of intervention.

Methods:

Selection: Seventy persons with diagnosis of RA and fatigue over 50 (0-100) will be recruited from the rheumatology clinic at Sahlgrenska University Hospital. Participants are randomized to an intervention group or a waiting list control group.

Intervention: The 12-week intervention period begins with an individual person-centered meeting to develop an individualized feasible self-care plan for the participant with extra focus on health-enhancing physical activity, stress management (relaxation exercise training and modified mindfulness techniques) and balance in daily life. A written consent, aiming to increase coherence, is signed. The participants will be asked to keep a journal about their strategies and reflections. Follow up meetings and contacts will be planned according to personal preferences.

Procedure: The participants are invited to a clinical examination before and after the 12-week intervention and at 6-month follow-up, assessing demographic data, disease activity, inflammation parameters, physical capacity and questionnaires of health status in RA. Primary outcome are questionnaires of single item- and multidimensional fatigue.

Analysis: Effects of the interventions will be analyzed using non-parametric statistics for between-group changes over time. Within-group changes over time will be analyzed for each group.

Expected results. New knowledge of fatigue is of importance for improvement of overall health of people with RA, as fatigue influences all aspects of their life, both private life and employment, thus decreasing the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* aging 20-65 years, disease duration >3 year, stable pharmacological treatment

Exclusion Criteria:

* Other serious physical or mental illness, lack of knowledge in Swedish language making answering the questionnaires impossible.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-10-10 (Actual); Study Completion 2014-10-10 (Actual)

PRIMARY OUTCOMES:
fatigue | 6months
  questionnaire

SECONDARY OUTCOMES:
Pain during previous week | 6months
  VAS
Physical function | 6months
  Performance based test
Disease activity | 6 months
  DAS-28
Health-related quality of life | 6 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa Mannerkorpi, Ass prof, Principal Investigator — Göteborg University, Dept of Rheumatology
Locations (1):
- rheumatology clinic at Sahlgrenska University Hospital, Gothenburg, Sweden